CLINICAL TRIAL: NCT00820612
Title: A Prospective, Randomized, Controlled Trial of Rectal Indomethacin in the Prevention of Post-ERCP Pancreatitis in High Risk Patients.
Brief Title: Rectal Indomethacin in the Prevention of Post-endoscopic Retrograde Cholangiopancreatography (ERCP) Pancreatitis in High Risk Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped by DSMB for overwhelming benefit of indomethacin (unethical to withhold indomethacin from patients)
Sponsor: University of Michigan (Other)
Collaborators: Indiana University School of Medicine (Other); University of Kentucky (Other); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Badih Joseph Elmunzer, Assistant Professor, Gastroenterology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HUM00022847
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Post-ERCP Pancreatitis
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Indomethacin suppository
  Interventions: Drug: Indomethacin
- 2 (Placebo Comparator): Placebo suppository
  Interventions: Other: Placebo suppositories

INTERVENTIONS:
Drug: Indomethacin — 100 mg PR once at the time of ERCP
  Arms: 1
Other: Placebo suppositories — 2 placebo suppositories at the time of ERCP
  Arms: 2

SUMMARY:
Pancreatitis (inflammation of the pancreas) is the most common complication of endoscopic retrograde cholangiopancreatography (ERCP), a procedure for the diagnosis and treatment of disorders of the pancreas and bile duct.

Preliminary data has shown that non-steroidal antiinflammatory drugs, when administered rectally, can reduce the risk of pancreatitis after ERCP. This study is intended to definitively determine whether rectally administered indomethacin (a non-steroidal antiinflammatory drug)is effective at preventing pancreatitis after ERCP.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, placebo-controlled, double-blinded clinical trial of rectal indomethacin in the prevention of post-ERCP pancreatitis in high risk patients.

ELIGIBILITY:
Inclusion Criteria:

Included patients are those undergoing ERCP and have one of the following:

1. Clinical suspicion of sphincter of Oddi dysfunction
2. History of post-ERCP pancreatitis (at least one episode)
3. Pancreatic sphincterotomy
4. Pre-cut (access) sphincterotomy
5. > 8 cannulation attempts
6. Pneumatic dilation of intact biliary sphincter
7. Ampullectomy

or at least 2 of the following:

1. Age < 50 years old & female gender
2. History of recurrent pancreatitis (at least 2 episodes)
3. ≥3 pancreatic injections, with at least one injection to tail
4. Pancreatic acinarization
5. Pancreatic brush cytology

Exclusion Criteria:

1. Unwillingness or inability to consent for the study
2. Age < 18 years
3. Intrauterine pregnancy
4. Breast feeding mother
5. Standard contraindications to ERCP
6. Allergy to Aspirin or NSAIDs
7. Renal failure (Cr > 1.4)
8. Active or recent (within 4 weeks) gastrointestinal hemorrhage
9. Acute pancreatitis (lipase peak) within 72 hours
10. Known chronic calcific pancreatitis
11. Pancreatic head malignancy
12. Procedure performed on major papilla/ventral panc duct in pt with pancreas divisum (no manipulation of minor papilla)
13. ERCP for biliary stent removal or exchange without anticipated pancreatogram
14. Subjects with prior biliary sphincterotomy now scheduled for repeat biliary therapy without anticipated pancreatogram
15. Anticipated inability to follow protocol
16. Endoscopist discretion: low risk (<10%) of post-ERCP pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Badih J Elmunzer, MD, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - University Hospitals Case Medical Center, Cleveland, Ohio

REFERENCES:
- [Derived] Elmunzer BJ, Scheiman JM, Lehman GA, Chak A, Mosler P, Higgins PD, Hayward RA, Romagnuolo J, Elta GH, Sherman S, Waljee AK, Repaka A, Atkinson MR, Cote GA, Kwon RS, McHenry L, Piraka CR, Wamsteker EJ, Watkins JL, Korsnes SJ, Schmidt SE, Turner SM, Nicholson S, Fogel EL; U.S. Cooperative for Outcomes Research in Endoscopy (USCORE). A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. N Engl J Med. 2012 Apr 12;366(15):1414-22. doi: 10.1056/NEJMoa1111103. PMID 22494121

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2009 and July 2011, 602 subjects were enrolled at 4 university-affiliated medical centers in the United States.
Pre-assignment Details: Of the 799 consented subjects, 169 were not randomized because an inclusion criterion was not met, 11 were not randomized because an exclusion criterion was met, and 17 were not randomized because ERCP not performed.
Groups:
- Placebo: 2 placebo suppositories. The suppositories were administered immediately after ERCP while the patient was still in the procedure room.
- Indomethacin: 2 50-mg indomethacin suppositories. The suppositories were administered immediately after ERCP while the patient was still in the procedure room.
Period: Overall Study
Arm/Group | Placebo | Indomethacin
Started | 307 | 295
Completed | 307 | 295
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Indomethacin | Total
Number analyzed (Participants) | 307 | 295 | 602
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 280 | 272 | 552
  >=65 years | 27 | 23 | 50
Age Continuous [Mean (Standard Deviation); unit: years] | 46.0 (13.1) | 44.5 (13.5) | 45.3 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 229 | 476
  Male | 60 | 66 | 126
Region of Enrollment [Number; unit: participants]
  United States | 307 | 295 | 602

OUTCOME MEASURES:

1. Primary Outcome: Post-ERCP Pancreatitis
Description: Subjects were diagnosed with post-ERCP pancreatitis if they experienced new upper abdominal pain, pancreatic enzyme elevation at least three times the upper limit of normal 24 hours after the procedure, and hospitalization of at least two nights.
Time Frame: 5 days
Population: 100% completed follow-up
Measure: Number; unit: participants
Arm/Group | Placebo | Indomethacin
Number analyzed (Participants) | 307 | 295
participants | 52 (37.6) | 27 (28.9)

ADVERSE EVENTS:
Time Frame: 30 days
Description: All reported adverse events were events potentially related to the study medication. The other major adverse event was post-ERCP pancreatitis, which was reported as the primary outcome, but would not be related to the treatment. All patients were systematically followed for adverse events.
Arm/Group | Placebo | Indomethacin
Serious Adverse Events (participants affected / at risk) | 61/307 | 31/295
Other Adverse Events (participants affected / at risk) | 0/307 | 0/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=307) | Indomethacin (N=295)
GI bleeding (Gastrointestinal disorders) | 7 (7) | 4 (4)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Post-ercp pancreatitis (Gastrointestinal disorders) | 52 (52) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No